CLINICAL TRIAL: NCT01740700
Title: Zenith® p-Branch® Multicenter Study
Brief Title: Zenith® p-Branch® OTS Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 12-002
Record Dates: First submitted 2012-10-19; First posted 2012-12-04 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Abdominal aortic aneurysm; Endovascular; Fenestration; Juxtarenal; Off-the-shelf; Pararenal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- p-Branch® (Experimental)
  Interventions: Device: p-Branch®

INTERVENTIONS:
Device: p-Branch® — Instead of making a large incision in the abdomen, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.
  Other Names: Endovascular graft; Endovascular stent; Stent-graft

SUMMARY:
The purpose of the Zenith® p-Branch® OTS Multicenter Study is to provide an early clinical experience and evaluate the safety and effectiveness of the Zenith® p-Branch® in the treatment of pararenal or juxtarenal abdominal aortic aneurysms (AAA).

ELIGIBILITY:
Inclusion Criteria:

* Pararenal or juxtarenal AAA ≥5.0 cm in diameter or 2 times the normal aortic diameter
* Pararenal or juxtarenal AAA with history of growth ≥0.5 cm/year
* Saccular aneurysm with aortic diameter greater than 1.5 times the normal aortic diameter that is deemed to be at risk for rupture based upon physician interpretation

Exclusion Criteria:

* Age <18 years
* Life expectancy <2 years
* Pregnant, breast-feeding, or planning on becoming pregnant within 60 months
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Unwilling or unable to comply with the follow-up schedule
* Simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study.)
* Additional medical restrictions as specified in the Clinical Investigation Plan
* Additional anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Technical success | Within 30 days
  Technical success is defined as successful access and deployment of the graft and patency of the vessels targeted by fenestrations.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Farber, MD, Principal Investigator — University of North Carolina
Locations (10):
- United States (10):
  - University of Florida, Gainesville, Florida
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Attaran RR, Bhalla A, Mena-Hurtado CI, Ochoa Chaar CI. Correlation between great saphenous length of treatment zone and diameter with improvement in symptoms after ablation. J Vasc Surg Venous Lymphat Disord. 2021 Nov;9(6):1443-1450. doi: 10.1016/j.jvsv.2021.02.013. Epub 2021 Mar 9. PMID 33706000
- [Derived] Farber MA, Oderich GS, Timaran C, Sanchez LA, Dawson Z; Zenith p-Branch Feasibility Study Investigators. Results from a prospective multicenter feasibility study of Zenith p-Branch stent graft. J Vasc Surg. 2019 Nov;70(5):1409-1418.e3. doi: 10.1016/j.jvs.2019.03.026. Epub 2019 Jun 27. PMID 31255472
- [Derived] Timaran DE, Knowles M, Ali T, Timaran CH. Fenestrated endovascular aneurysm repair among octogenarians at high and standard risk for open repair. J Vasc Surg. 2017 Aug;66(2):354-359. doi: 10.1016/j.jvs.2016.11.064. Epub 2017 Feb 16. PMID 28216359